CLINICAL TRIAL: NCT02144129
Title: Effects of Different Types of Whole Body Electromyostimulation (WB-EMS) Application on Body Composition, Muscle Strength and Quality of Life in Patients With Ulcerative Colitis
Brief Title: Effects of WB-EMS in Ulcerative Colitis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Professor Dr., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS_COL; Substudy 1 (Other: Medizinische Klinik 1, University of Erlangen-Nurnberg)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Ulcerative Colitis
Keywords: Whole Body Electromyostimulation; Inflammatory Bowel Disease; Lean Body Mass; Muscle Strength
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- active WB-EMS (Experimental): 2 sessions/week with 20 min of active WB-EMS application
  Interventions: Other: active Whole Body Electromyostimulation; Device: WB-EMS application
- Passive WB-EMS (Experimental): 2 sessions/week with 20 min of passive WB-EMS application in a resting supine position
  Interventions: Other: Passive WB-EMS
- Inactive Control Group (No Intervention): sedentary non-training control group

INTERVENTIONS:
Other: active Whole Body Electromyostimulation
  Arms: active WB-EMS
Other: Passive WB-EMS
  Arms: Passive WB-EMS
Device: WB-EMS application
  Arms: active WB-EMS

SUMMARY:
The purpose of this study is to determine the effect of 12 weeks of WB-EMS either applicated passive in a supine resting position or active during slight movements compared with a non-training control group on body composition, muscle strength and QoL in patients with ulcerative colitis.

Our main hypothesis is that active WB-EMS application is significantly more favorable to address our primary endpoints compared with passive application.

Our secondary hypothesis is that passive WB-EMS application is significantly more favorable to address our primary endpoints compared with non-training control.

ELIGIBILITY:
Inclusion Criteria:

* ulcerative colitis
* ambulatory subjects

Exclusion Criteria:

* variables that conflicts with WB-EMS application (e.g. cardiac pacemakers)
* absence of more than two weeks during the interventional period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Lean Body Mass | 12 weeks, baseline to 12 week follow-up
  Lean Body Mass (LBM) and Appendicular Skeletal Muscle Mass (ASMM) as assessed by Dual-Energy-x-Ray Absorptiometry (DXA)
Isokinetic muscle strength | 12 weeks, baseline to 12 week follow-up
  Isokinetic muscle strength of the leg extensors and - flexors as assessed by a isokinetic leg strength

SECONDARY OUTCOMES:
Quality of Life (QoL) | 12 weeks, baseline to 12 week follow-up
  QoL as assessed by inflammatory bowel disease questionnaire (IBDQ-D) and Depression Scores
Isometric muscle strength | 12 weeks, baseline 12 week follow-up
  Isometric strength of the trunk flexors.

OTHER OUTCOMES:
Aerobic capacity | 12 weeks, baseline to 12 weel follow-up
  Aerobic capacity as assessed by 6 min walking test
Inflammatory Markers | 12 weeks, baseline to 12 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül Zopf, MD, Study Chair — University of Erlangen-Nürnberg; Wolfgang K Kemmler, PhD, Study Director — University of Erlangen-Nürnberg Medical School; Michael Weineck, MS, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Medizinische Klinik 1, University of Erlangen-Nurnberg, Erlangen, Franconia, Germany

REFERENCES:
- [Background] Kemmler W, von Stengel S. Whole-body electromyostimulation as a means to impact muscle mass and abdominal body fat in lean, sedentary, older female adults: subanalysis of the TEST-III trial. Clin Interv Aging. 2013;8:1353-64. doi: 10.2147/CIA.S52337. Epub 2013 Oct 7. PMID 24130433
- [Background] Kemmler W, Bebenek M, Engelke K, von Stengel S. Impact of whole-body electromyostimulation on body composition in elderly women at risk for sarcopenia: the Training and ElectroStimulation Trial (TEST-III). Age (Dordr). 2014 Feb;36(1):395-406. doi: 10.1007/s11357-013-9575-2. Epub 2013 Aug 16. PMID 23949160